CLINICAL TRIAL: NCT06942923
Title: A Phase I, Randomised, Investigator- and Participant-blinded, Placebo-Controlled, Study to Assess the Safety, Tolerability, and Pharmacodynamics of AZD4144 in Participants With Obesity
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacodynamics of AZD4144 in Participants With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D9441C00004
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants
Keywords: Cardiorenal disease; Atherosclerotic cardiovascular disease; Chronic kidney disease; Type 2 Diabetes Mellitus; Atherosclerosis; Obesity
MeSH Terms: conditions — Atherosclerosis; Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD4144 (Experimental): Participants will receive a single oral dose of AZD4144 under fasted conditions once daily for 28 days.
  Interventions: Drug: AZD4144
- Placebo (Placebo Comparator): Participants will receive a single oral dose of matching placebo to AZD4144 under fasted conditions once daily for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4144 — AZD4144 will be administered orally as per arms they have been assigned.
  Arms: AZD4144
Drug: Placebo — Placebo will be administered orally as per arms they have been assigned.
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the safety and tolerability, and pharmacodynamics (PD) of AZD4144 administered as repeated daily oral dosing.

DETAILED DESCRIPTION:
This is placebo-controlled, parallel group and single centre study in healthy male and female participants with obesity and no known Atherosclerotic cardiovascular disease (ASCVD), chronic kidney disease (CKD), or Type 2 Diabetes Mellitus.

Participants will be randomized in the ratio of 1:1 to receive either AZD4144 or placebo.

This study will comprise of:

* A screening period of 28 days.
* The treatment duration will be up to 28 days.
* The visit frequency will be weekly up to a Follow-up Visit, followed by a Final Follow-up Visit 28 days after the final dose of AZD4144.

ELIGIBILITY:
Key Inclusion Criteria:

* Serum hsCRP > 2 milligrams per liter (mg/L).
* All females must have a negative pregnancy test at the Screening Visit and at the randomization visit (Visit 2).
* Females of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception to avoid pregnancy from the time of first administration of study intervention until 3 months after the Final Follow-up Visit.
* Have a body mass index (BMI) greater than or equal to (≥) 30 and less than or equal to (≤) 45 kilograms per meter^2 (kg/m^2).

Key Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History of Myocardial infarction (MI), coronary revascularisation, stroke, revascularisation for peripheral arterial disease, or other pre-existing Cardiovascular (CV) diseases.
* History of Diabetes (Type 1 and Type 2) or glycated haemoglobin (HbA1c) ≥6.5%.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Any skin disorder, history of, or ongoing clinically significant allergy/hypersensitivity.
* Clinically significant serious active and chronic infections within 60 days prior to randomization.
* Known history of primary immunodeficiency (congenital or acquired) or an underlying condition that predisposes to infection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | From Screening (Day -28 to Day -2) to final follow-up (Day 56)
  The safety and tolerability of AZD4144 compared with placebo will be assessed.
Relative change from baseline in systemic interleukin-6 (IL-6) levels | From baseline to 4 weeks
  The effect of AZD4144 on circulating inflammatory biomarker IL-6 compared with placebo will be assessed.

SECONDARY OUTCOMES:
Relative change from baseline in systemic IL-18 levels | From baseline to 4 weeks
  The effect of AZD4144 compared with placebo on circulating biomarker IL-18 will be assessed.
Relative change from baseline in high-sensitivity C-reactive protein (hsCRP) levels | From baseline to 4 weeks
  The effect of AZD4144 compared with placebo on circulating biomarker hsCRP will be assessed.
Observed lowest concentration before the next dose is administered (Ctrough) of AZD4144 | From Day 1 to Day 28
  The pharmacokinetics (PK) of AZD4144 in participants with obesity will be assessed.
Maximum observed drug concentration (Cmax) of AZD4144 | From Day 1 to Day 28
  The PK of AZD4144 in participants with obesity will be assessed.
Time to reach maximum observed concentration (tmax) of AZD4144 | From Day 1 to Day 28
  The PK of AZD4144 in participants with obesity will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST /Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/